CLINICAL TRIAL: NCT05169840
Title: Genetic Risk Stratification for Primary Prevention of CAD in Men and Pre & Post-menopausal Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Chandler Regional Medical Center (Unknown); Mercy Gilbert Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19-500-384-50-17
Record Dates: First submitted 2021-05-13; First posted 2021-12-27 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Genetic Predisposition to Disease
Keywords: Genetic Risk Score; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Genetic Predisposition to Disease; Genetic Risk Score

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collected in a PAXgene tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Genetic Risk Score for Coronary Artery Disease — Blood samples will be genotyped for million of genetic risk variants for Coronary Artery Disease (CAD)
  Other Names: Conventional Risk Score for Coronary Artery Disease

SUMMARY:
The investigators propose to genotype males and females at age 40 years and older, who are asymptomatic and without known heart disease (N=2000). DNA from a blood sample will be genotyped for millions of genetic risk variants for CAD by Baylor College of Medicine Human Genome Sequencing Center Clinical Laboratory (HGSC-CL) in a CLIA-approved laboratory.

The overall objective after 2 years is to determine if genetic screening for risk of CAD in asymptomatic men and women has the discriminatory power to detect those at highest risk who would potentially benefit most from appropriate primary prevention. It will also determine whether the GRS is appropriate for different ethnic and race groups such as Hispanics, African Americans and Whites, and to what extent those individuals knowing that they are at higher risk, are more likely to seek further advice on management of the risks (either through changes in lifestyle or therapy).

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is an epidemic, being the most common cause of death in the world. CAD is preventable as shown by clinical trials that reduce conventional risk factors such as hypercholesterolemia. Epidemiologists have claimed 40-60% of pre-disposition to CAD is genetic. In 2007, the investigators and the Icelandic group independently identified the first genetic risk variant for CAD, 9p21. Through the formation of an international consortium, the investigators have now identified over 200 genetic risk variants predisposing to CAD. Utilizing a genetic risk score (GRS) based on these variants for CAD, several studies have retrospectively documented the risk stratification for primary or secondary prevention of CAD to be superior and relatively independent of, conventional risk factors. Studies in over 1 million individuals show those with the highest genetic risk exhibit up to a 4-fold increased risk of CAD. More importantly, those with a high GRS and a more favorable lifestyle experienced 50% reduction in cardiac events. In the high risk group one needs to treat only 13 individuals with statin therapy to prevent one cardiac event. The GRS detects those at high risk who will benefit most from primary prevention. The myth that one cannot treat genetic predisposition has been dispelled. While secondary prevention of CAD has been successful, application of primary prevention has until now lacked a risk marker to detect those who would benefit most. Given only 47% of the population will experience a cardiac event, administering preventive therapy, such as statin, to everyone would be unnecessarily expensive and inappropriate. Since the GRS is determined at birth, and does not change during one lifetime it is close to ideal for primary prevention. GRS detects among asymptomatic individuals at any age those at high-risk for CAD, who will benefit most from preventive therapy.

The investigators propose to genotype males and females at age 40 years and older, who are asymptomatic and without known heart disease (N=2000). DNA from a blood sample will be genotyped for millions of genetic risk variants for CAD by Baylor College of Medicine Human Genome Sequencing Center Clinical Laboratory (HGSC-CL) in CLIA-approved laboratories.

The derived GRS will be added to the conventional risk score using the American College of Cardiology/American Heart Association's (AHA) Pooled Cohort Atherosclerotic Cardiovascular Disease (ASCVD) Risk Equation. In the female cohort, investigators will also be screening for female-specific risk factors that have been added to the ACC/AHA 2018 Blood Cholesterol Guidelines to be used as risk enhancers. Everyone at high risk, will be referred to their physician for further management and given the opportunity for genetic counseling by a member of the research team. Completion of the 2 year recruitment will meet the objectives, however, an annual follow-up will be obtained by electronic survey via REDCap, letter or phone call over a 10 year period as it may provide information on long term genetic prediction.

The overall objective after 2 years is to determine if genetic screening for risk of CAD in asymptomatic men and women has the discriminatory power to detect those at highest risk who would potentially benefit most from appropriate primary prevention. It will also determine whether the GRS is appropriate for different ethnic and race groups such as Hispanics, African Americans and Whites, and to what extent those individuals knowing that they are at higher risk, are more likely to seek further advice on management of the risks (either through changes in lifestyle or therapy). The investigators expect to complete recruitment in two years and prove that the GRS is appropriate for clinical application and can detect individuals that have a 50% or more increase in risk for CAD.

ELIGIBILITY:
Inclusion Criteria:

* Males 40 to 60 years of age
* Females 40 to 60 years of age
* No known cardiovascular disease
* Willing and able to sign consent

Exclusion Criteria:

* Prisoners
* Prior percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
* Known ischemia on non-invasive testing
* Ischemic cerebrovascular event
* Peripheral arterial disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People 40 to 60 years old who are asymptomatic and without known heart disease.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Genetic Risk Score (GRS) | 2 years
  The GRS will be calculated by summing the product of the number of risk variants inherited by each individual times their associated Coronary Artery Disease risk. The score will be classified into low, intermediate and high.
Participant's response on the informed consent regarding their wish to learn about their genetic risk. | 2 years
  Participants will be asked on the informed consent whether they would like to learn about their calculated genetic risk and will provide a yes or no answer.
Spread of the Genetic Risk Score (GRS) in Hispanics or African Americans vs those of European descent. | 2 years
  Since previous studies utilizing the GRS have been predominately in white individuals of European descent data will be stratified to determine if the GRS has the same risk stratification power in Hispanics and African Americans vs those of European descent.
Percentage of participants with a high Genetic Risk Score (GRS) who take action as a result. | 10 years
  Participants with a high GRS will be asked at follow up whether they have followed through on recommendations to seek further care, started any new therapies and/or if they have made lifestyle changes as a result. This will be assessed annually for 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Roberts, MD, Principal Investigator — Dignity Health
Locations (3):
- United States (3):
  - Chandler Regional Medical Center, Chandler, Arizona
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - St Joseph's Hospital and Medical Center, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No